CLINICAL TRIAL: NCT01804790
Title: Randomized Phase III Study Comparing Preoperative Chemoradiotherapy Alone Versus Neoadjuvant Chemotherapy With Folfirinox Regimen Followed by Preoperative Chemoradiotherapy for Patients With Resectable Locally Advanced Rectal Cancer
Brief Title: Efficacy of Neoadjuvant Folfirinox Regimen in Patients With Resectable Locally Advanced Rectal Cancer
Acronym: Néofirinox
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 23 - UCGI 23; 2011-004406-25 (EudraCT Number)
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cancer of the Rectum
Keywords: rectum; cancer; locally advanced
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : Radiotherapy + capecitabine (Active Comparator): Chemoradiotherapy 5 weeks (50 Grays (Gy), 2 Gy/session ; 25 fractions) + capecitabine 800 mg/m² twice daily 5 days/7, excluding weekends), then 6-8 weeks after chemoradiation, surgery with total mesorectal excision (TME), followed by adjuvant chemotherapy for 6 months, either mFolfox6 or capecitabine, depending on the center's choice.
  Interventions: Radiation: Radiotherapy 50 Gy; Drug: Capecitabine; Procedure: TME surgery; Drug: mFolfox6 or capecitabine
- Arm B : Chemotherapy then radiochemotherapy (Experimental): Drug: Chemotherapy mFolfirinox
  Investigational arm: Neoadjuvant CT mFolfirinox, 6 cycles (ca. 3 months; each cycle = 2 weeks):
  oxaliplatin: 85 mg/m² in 2 hours at D1 irinotecan: 180 mg/m² in 90 min at D1 folinic acid: 400 mg/m² simultaneously in 2 hours at D1 during the irinotecan infusion 5-fluorouracil (5-FU): 2400 mg/m² continuous infusion during 48 hours (1200 mg/m² at D1 and D2), every 14 days during 2 months (4 cycles).
  Then followed by 5 weeks of chemoradiotherapy 50 Gy (2 Gy/session, 5 sessions per week) + capecitabine 800 mg/m² twice daily 5 days/7), then surgery with TME 6-8 weeks after chemoradiation, followed by 3 months of adjuvant chemotherapy, either mFolfox6 or capecitabine depending on the center's choice.
  Interventions: Drug: mFolfirinox; Radiation: Radiotherapy 50 Gy; Drug: Capecitabine; Procedure: TME surgery; Drug: mFolfox6 or capecitabine

INTERVENTIONS:
Drug: mFolfirinox — Investigational arm: Neoadjuvant chemotherapy mFolfirinox, 4 cycles: oxaliplatin: 85 mg/m² in 2 hours at D1 irinotecan: 180 mg/m² in 90 min at D1 folinic acid: 400 mg/m² simultaneously in 2 hours at D1 during the irinotecan infusion 5-FU: 2400 mg/m² continuous infusion during 48 hours (1200 mg/m² at D1 and D2), every 14 days during 2 months (4 cycles), then CRT (50 Gy (2 Gy/session, 25 fractions) + capecitabine 800 mg/m² twice a day 5 days/7), then surgery with TME 6-8 weeks after chemoradiation, and 4 months of adjuvant CT depending on the center's choice.
  Arms: Arm B : Chemotherapy then radiochemotherapy
Radiation: Radiotherapy 50 Gy — 5 radiations per week of 2 Gy for 5 weeks
Drug: Capecitabine — 1600 mg/m² (800 mg/m² twice daily) for 5 weeks
Procedure: TME surgery
Drug: mFolfox6 or capecitabine — oxaliplatine 85 mg/m² (day 1 of cycle; perfusion in 2h), folinic acid 400 mg/m² (day 1 of cycle perfusion in 2h), 5-FU (bolus 400 mg/m² in 10 min and 2400 mg/m² perfusion continuous 46h). Arm A - 12 cycles ; Arm B - 6 cycles OR Capecitabine 2500 mg/m²/day (Each cycle consists of 1250 mg/m² twice daily for D1-14 then pause therapeutic from D15-21). Arm A - 8 cycles; Arm B 4 cycles.

SUMMARY:
National, multi-center, open-label,randomized, 2-arm phase III superiority trial, comparing neoadjuvant chemotherapy (CT) with mFolfirinox followed by preoperative chemoradiotherapy (CRT), versus preoperative CRT in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
Methodology This is a biomedical research, national, multicenter, open-label randomized, 2-arm phase III superiority trial, comparing neoadjuvant CT with mFolfirinox then preoperative CRT, versus immediate preoperative CRT, in patients with locally advanced rectal cancer Randomized Phase III study with stopping rules Stratification : center, gender, tumor location in the rectum (<6 cm from anal verge versus ≥6 cm), initial stage (cT3 vs cT4, and cN0 vs cN+)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven rectal adenocarcinoma
* Stages cT3 with risk of local recurrence or cT4, M0 and for which a multidisciplinary meeting recommend preoperative CRT
* Resectable tumor, or considered as potentially resectable after CRT
* No distant metastases
* Patient eligible for surgery
* Patient aged from 18 to 75 years
* World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status 0/2.
* No heart failure or coronary heart disease symptoms (even controlled).
* No peripheral neuropathy > grade 1
* No prior radiotherapy of the pelvis for any reason and no previous CT
* No major comorbidity that may preclude the delivery of treatment and no active infection (HIV or chronic hepatitis B or C).
* Adequate contraception in fertile patients.
* Adequate hematologic function
* Adequate hepatic function
* Signed written informed consent

Exclusion Criteria:

* Metastatic disease
* Unresectable rectal cancer, including prostatic involvement or extension to pelvic floor muscles
* Contraindication to 5-FU, or to oxaliplatin or to irinotecan, including Gilbert disease or genotype UGT1A1
* Medical history of chronic diarrhea or inflammatory disease of the colon or rectum
* Medical history of angina pectoris or myocardial infarction
* Progressive active infection or any other severe medical condition that could jeopardize treatment administration
* Other concomitant cancer, or medical history of cancer other than treated in situ cervical carcinoma or basocellular carcinoma or spinocellular carcinoma
* Patient included in another clinical trial testing an investigational agent.
* Pregnant or breast-feeding woman.
* Persons deprived of liberty or under guardianship or incapable of giving consent
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 3 years
  To compare the 3-year disease-free survival between the investigational arm and the control arm.

SECONDARY OUTCOMES:
Overall survival | 7 years
  Overall survival will be defined as the time from randomisation to the time of occurrence of the first death regardless to its cause. Patients alive at the time of analysis will be censored at the date of the last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry CONROY, PROF, Principal Investigator — centre Alexis Vautrin les Nancy
Locations (36):
- France (36):
  - Centre hospitalier Universitaire d'Amiens, Amiens
  - ICO - Site Paul Papin, Angers
  - Centre hospitalier d'Auxerre, Auxerre
  - Centre Hospitalier de Beauvais, Beauvais
  - Institut de Cancérologie de Franche Comté, Besançon
  - Centre Hospitalier de Blois, Blois
  - Hopital Avicenne, Bobigny
  - Clinique Tivoli, Bordeaux
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Chd de La Roche Sur Yon - Les Oudairies, La Roche-sur-Yon
  - Centre Bourgogne, Lille
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hopital Prive Jean Mermoz, Lyon
  - Ap Hm - Hopital de La Timone - Adultes, Marseille
  - Institut de Cancérologie de Franche Comté, Montbéliard
  - Centre Azuréen de cancérologie, Mougins
  - Hopital Emile Muller, Mulhouse
  - centre Alexis Vautrin, Nancy
  - Polyclinique de Gentilly, Nancy
  - Centre Antoine Lacassagne, Nice
  - Groupe Hospitalier La Pitie-Salpetriere, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Regional D'Annecy, Pringy
  - Hopital Robert Debre, Reims
  - Institut Jean Godinot, Reims
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Hopital Saint Gregoire, Saint-Grégoire
  - ICO - Site René Gauducheau, Saint-Herblain
  - Clinique Mutualiste de L'Estuaire, Saint-Nazaire
  - Centre Hospitalier de la Réunion - Site du GHSR, Saint-Pierre
  - Centre Paul Strauss, Strasbourg
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.

REFERENCES:
- [Result] Conroy T, Bosset JF, Etienne PL, Rio E, Francois E, Mesgouez-Nebout N, Vendrely V, Artignan X, Bouche O, Gargot D, Boige V, Bonichon-Lamichhane N, Louvet C, Morand C, de la Fouchardiere C, Lamfichekh N, Juzyna B, Jouffroy-Zeller C, Rullier E, Marchal F, Gourgou S, Castan F, Borg C; Unicancer Gastrointestinal Group and Partenariat de Recherche en Oncologie Digestive (PRODIGE) Group. Neoadjuvant chemotherapy with FOLFIRINOX and preoperative chemoradiotherapy for patients with locally advanced rectal cancer (UNICANCER-PRODIGE 23): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2021 May;22(5):702-715. doi: 10.1016/S1470-2045(21)00079-6. Epub 2021 Apr 13. PMID 33862000
- See also: Lancet Oncology 2021 Apr 13: publication of results — https://pubmed.ncbi.nlm.nih.gov/33862000/